CLINICAL TRIAL: NCT04394975
Title: A Phase III, Randomized, Open-label, Active Controlled, Multicenter Study on Toripalimab Combined With Axitinib Versus Sunitinib Monotheraphy as a First-Line Treatment for Unresectable or Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Study to Evaluate the Efficacy and Safety of Toripalimab in Combination With Axitinib Versus Sunitinib Monotherapy in Advanced Renal Cell Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS001-036-Ⅲ-RCC
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Primary Disease: Unresectable or Metastatic Renal Cell Carcinoma Focus of the Study:PFS Assessed by IRC Per RECIST 1.1
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Toripalimab+axitinib combination therapy. Participants receive Toripalimab 240mg intravenously every 3 weeks plus axitinib 5mg orraly twice daily.
  Interventions: Combination Product: Biological : Toripalimab Drug: Axitinib
- Control group (Active Comparator): Sunitinib monotherapy. Participants receive sunitinib 50mg orally once daily for 4 weeks and then are off treatent for 2 weeks, or once daily for 2weeks and then are off treatent for 1 week.
  Interventions: Drug: sunitinib

INTERVENTIONS:
Combination Product: Biological : Toripalimab Drug: Axitinib — Biological: Toripalimab, Intravenous infusion Drug: Axitinib, oral tablet
  Arms: Test group
Drug: sunitinib — Drug: Sunitinib, oral capsule
  Arms: Control group

SUMMARY:
This is a randomized, open-label, controlled, multicenter, phase III trial to compare the efficacy and safety of Toripalimab in combination with axitinib to sunitinib monotherapy as a first-line therapy for advanced RCC. Eligible patients will be randomized 1:1 to receive the combination therapy of Toripalimab and axitinib or sunitinib monotherapy.

ELIGIBILITY:
Inclusion criteria:

1. Fully understand and be willing to provide written informed consent.
2. Male or female with age ≥ 18 years and <80 years.
3. Have received no prior systemic therapy after previous metastasis for RCC, histologically confirmed diagnosis of unresectable, recurrent or metastatic RCC with clear cell component with or without sarcomatoid features,Prior cytokine therapy was allowed.
4. The IDMC score was medium to high risk.
5. Having at least one measurable disease per RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if re-progression has been demonstrated.
6. Provide archival tumor tissues or newly obtained biopsies if patients participate in the exploratory study.
7. ECOG PS 0 or 1.
8. Adequate function of vital organs:

Bone marrow function (without blood or blood products transfusion, without hematopoietic stimulating factor or other medication to improve blood cell count within 2 days prior to first dose of study drug):

Absolute neutrophil count (ANC) ≥ 1.5×109/L. Platelets ≥ 100×109/L. Hemoglobin ≥ 9.0g/dL or ≥ 5.6mmol/L.

Renal function:

Serum creatinine ≤ 1.5×ULN

Hepatic function:

Serum total bilirubin ≤1.5×ULN or total bilirubin levels >1.5×ULN with direct bilirubin ≤ ULN. AST and ALT ≤2.5 × ULN, ≤5×ULN in those with hepatic metastasis.

Endocrine function:

Normal thyroid stimulating hormone, or abnormal TSH whilst normal FT3 and FT4.

Coagulation function:

International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN, and activated partial thromboplastin time (aPTT) ≤1.5×ULN, Subjects receiving anticoagulant therapy (e.g., heparin or warfarin) may participate in the study with PT or aPTT levels within the scope of the proposed therapy and monitored during study treatment.Left ventricular ejection fraction (LVEF) ≥ 50%.

8. Being willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

10. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first treatment dose. Female subjects of childbearing potential and male subjects whose partners are of childbearing potential must agree to use a highly effective methods of contraceptive throughout the study and for 180 days after the last dose of study therapy.

Exclusion criteria:Bone marrow functiPatients with any of the following conditions will not be included in the study:

1. PriorAnti-PD-1, PD-L1 or CTLA-4 agents ).
2. Prior systemic anti-cancer therapy after metastasis (e.g., VEGF/VEGFR or mTOR targeting agents, including (but not limited to) sunitinib, axitinib, sorafenib, pazopanib, cabozantinib, lenvatinib, bevacizumab or everolimus.
3. Progression or recurrence during neoadjuvant/adjuvant therapy for renal cell cancer or within 12 months after the last dose treatment.
4. Has participated or is currently participating in a trial of investigational agent within 4 weeks prior to the first dose of study treatment, unless observational (non-interventional) clinical study or follow-up period of interventional study.
5. Had major surgery (judged by investigators) within 4 weeks prior to the first dose of study treatment or has not recovered from prior surgery.
6. Has traditional Chinese medicine or Chinese patent medicine preparation with anti-cancer indication within 2 weeks prior to the first dose of study treatment.
7. Requiring corticosteroids (Prednisone >10 mg/day or equivalent analogue) or other immunosuppressive agents within 2 weeks prior to the first dose of study treatment. Patients without active autoimmune disease using inhaled prednisone >10 mg/day will not be excluded from the study.
8. Has a history of organ transplantation or required long-term treatment with corticosteroids.
9. Hypothyroidism, hypoadrenalism or hypopituitarism that can be controlled only with hormone replacement therapy, type I diabetes, psoriasis or leucoderma not requiring systematic treatment.
10. Not recovered from the toxicity of prior anti-cancer therapy, i.e., not recovered to baseline, Grade 0-1 (NCI-CTCAE 5.0, except alopecia) or per inclusion/exclusion criteria in protocol. Under rational expectation, irreversible toxicities (e.g., hearing loss) which will not be worsened by study treatments may be enrolled in the study.
11. Has an additional malignancy that has progressed or required treatment within 5 years prior to randomization (basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ such as breast cancer, prostate cancer are acceptable if they have undergone potentially curative therapy；Remarks: Localized low-risk prostate cancer [ patietns with stage ≤ T2a, Gleason score ≤ 6 and PSA < 10ng/mL at the time of diagnosis (as measured) can be included in this study if the subject has received radical therapy and has no evidence for biochemical recurrence(PROSTATE specific antigen,PSA)].
12. Has a history of active central nervous system (CNS) metastasis or CNS metastasis had been confirmed by radiological examination (MRI or CT) at baseline within 30 days prior to the first dose of study drug.Subjects may participate who had been stable at least for 3 months after prior surgery or RT for brain or meningeal metastasis and discontinued systemic treatment with corticosteroids (Prednisone >10 mg/day or equivalent analogue) for at least 4weeks. Subjects may participate in the study if their CNS metastases are adequately treated to meet the requirements specified in the inclusion criteria, and their neurological symptoms recover to grade 0-1 (CTCAE 5.0) for at least 2 weeks prior to inclusion (except for residual signs or symptoms associated with CNS treatment).
13. Poorly controlled hypertension (systolic blood pressure ≥ 150mmHg and/or diastolic blood pressure ≥ 90mmHg).
14. Presence of the following cardiovascular events within 6 months prior to randomization:

    1. Myocardial infarction
    2. Unstable angina pectoris
    3. Cardiac angioplasty or stent
    4. Coronary/peripheral artery bypass graft
    5. Grade III or IV congestive heart failure per New York Heart Association
    6. Cerebrovascular accident or transient ischemic attack
15. QT interval (QTc) ≥ 480 msec corrected with heart rate (Bazett's formula);
16. Has active hemorrhage or history of other significant hemorrhage episodes within 30 days prior to randomization.
17. Has deep vein thrombosis or pulmonary embolism within 6 months prior to randomization.
18. Has arterial thrombosis within 12 months prior to randomization.
19. Has clinically significant gastrointestinal (GI) abnormalities including:

    1. Malabsorption, total gastrectomy or any other condition that might affect the absorption of orally taken medication.
    2. Active ulcer under treatment in the past 6 months;
    3. Active GI bleeding (e.g., hematemesis, hematochezia or melena) in the past 3 months, and without evidence of resolution documented by endoscopy or colonoscopy.
    4. Intraluminal metastatic lesion with suspected hemorrhage, inflammatory bowel disease, ulcerative colitis, GI perforation, or other GI conditions associated with increased risk of perforation.
20. Has a history of or current (non-infective) pneumonia/ interstitial lung disease that required steroids.
21. Has an active infection requiring systemic therapy. Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV antibody positive), HBV or HCV infection (Patients with positive HBsAg or negative HBsAg, but positive HBcAb will be enrolled in the study when HBV DNA was tested in central laboratory and lower than ULN. Patients with a history of HCV infection may participate in the study if the result of HCV RNA test was negative during screening period).
22. Has received a live virus vaccine within 30 days prior to randomization, including (but not limited to) mumps, rubella, measles, varicella/ herpes zoster (chicken pox), yellow fever, rabies, Bacille Calmette-Guérin (BCG) and typhoid vaccine. Inactivated virus vaccines are allowed.
23. Has a history of hypersensitivity reaction, including (but not limited to) antibodies and TKIs.
24. Known history of psychiatric disorders or drug abuse.
25. Has evidence of inadequate wound healing.
26. Has current use (within 7 days of randomization) or anticipated need for treatment drugs what are known strong CYP3A4/5 inhibitor and CYP3A4/5 inducer (including, but not limited to, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin and St. John's wort) or the drugs that are known with proarrhythmic potential (including, but not limited to, terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol and benazapril, etc.).
27. Has a history or current evidence on any condition, therapy or laboratory abnormality that might confound the results of the study, interfere with subject's participation for the full duration of the study, or is not in the best interest of subject to participate, in the opinion of investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
PFS assessed by IRC per RECIST 1.1. | 3 years
  To compare the progression-free survival (PFS) per response evaluation criteria in solid tumors (RECIST) 1.1 as assessed by independent review committee (IRC) in subjects treated with Toripalimab plus axitinib vesus sunitinib monotherapy as a first-line treatment for advanced RCC.

SECONDARY OUTCOMES:
PFS assessed by investigators per RECIST 1.1; | 3 years
  The treatment effect of with Toripalimab plus axitinib vesus sunitinib monotherapy, will be assessed using RECIST 1.1 to determine tumor response;
ORR assessed by investigators and IRC per RECIST 1.1, respectively; | 3 years
  The treatment effect of with Toripalimab plus axitinib vesus sunitinib monotherapy, will be assessed using IRC and RECIST 1.1 to determine tumor response;
DOR, assessed by investigators and IRC per RECIST 1.1, respectively; | 3 years
  The treatment effect of with Toripalimab plus axitinib vesus sunitinib monotherapy, will be assessed using IRC and RECIST 1.1 to determine tumor response;
DCR assessed by investigators and IRC per RECIST 1.1, respectively; | 3 years
  The treatment effect of with Toripalimab plus axitinib vesus sunitinib monotherapy, will be assessed using IRC and RECIST 1.1 to determine tumor response;
overall survival rate assessed by investigators and IRC per RECIST 1.1, respectively; | 3 years
  The treatment effect of with Toripalimab plus axitinib vesus sunitinib monotherapy, will be assessed using IRC and RECIST 1.1 to determine tumor response;
OS assessed by investigators and IRC per RECIST 1.1, respectively; | 3 years
  The treatment effect of with Toripalimab plus axitinib vesus sunitinib monotherapy, will be assessed using IRC and RECIST 1.1 to determine tumor response;
Incidence and grade of AEs and SAEs per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, incidence of ≥ grade 3 AE; | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Incidence and grade of AEs and SAEs related to study drugs per NCI-CTCAE version 5.0, AEs ≥ grade 3 related to the study drugs. | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
Biomarker | 2 years
  Correlation between biomarker (PD-L1) and the efficacy of Toripalimab

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

REFERENCES:
- [Derived] Yan XQ, Ye MJ, Zou Q, Chen P, He ZS, Wu B, He DL, He CH, Xue XY, Ji ZG, Chen H, Zhang S, Liu YP, Zhang XD, Fu C, Xu DF, Qiu MX, Lv JJ, Huang J, Ren XB, Cheng Y, Qin WJ, Zhang X, Zhou FJ, Ma LL, Guo JM, Ding DG, Wei SZ, He Y, Guo HQ, Shi BK, Liu L, Liu F, Hu ZQ, Jin XM, Yang L, Zhu SX, Liu JH, Huang YH, Xu T, Liu B, Sun T, Wang ZJ, Jiang HW, Yu DX, Zhou AP, Jiang J, Luan GD, Jin CL, Xu J, Hu JX, Huang YR, Guo J, Zhai W, Sheng XN. Toripalimab plus axitinib versus sunitinib as first-line treatment for advanced renal cell carcinoma: RENOTORCH, a randomized, open-label, phase III study. Ann Oncol. 2024 Feb;35(2):190-199. doi: 10.1016/j.annonc.2023.09.3108. Epub 2023 Oct 21. PMID 37872020